CLINICAL TRIAL: NCT02738996
Title: Investigating the Response of Glycaemic Excursions in Type-2 Diabetes to Interrupting Prolonged Sedentary Behaviour (Sitting)
Brief Title: Role of Interrupting Sedentary Time in Management of Type-2 Diabetes
Acronym: Just_StandUp
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Glasgow Caledonian University (Other)
Collaborators: University of Strathclyde (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Just_StandUp
Record Dates: First submitted 2016-03-30; First posted 2016-04-14 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-03

CONDITIONS: Diabetes
Keywords: Diabetes; Sedentary Lifestyle
MeSH Terms: conditions — Diabetes Mellitus; Sedentary Behavior | interventions — Sitting Position

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- 60-30 min (Experimental): Sitting for 8 hours interrupted by 3 min of light intensity walking (LIW, 3.2 km/h) breaks every 60 min and 30 min
  Interventions: Behavioral: Sedentary time breaks either every 60 minutes; Behavioral: Sedentary time breaks either every 30 minutes
- 30-15 min (Experimental): Sitting for 8 hours interrupted by 3 min of light intensity walking (LIW, 3.2 km/h) breaks every 30 min and 15 min
  Interventions: Behavioral: Sedentary time breaks either every 30 minutes; Behavioral: Sedentary time breaks every 15 minutes
- 15-60 min (Experimental): Sitting for 8 hours interrupted by 3 min of light intensity walking (LIW, 3.2 km/h) breaks every 15 min and 60 min
  Interventions: Behavioral: Sedentary time breaks either every 60 minutes; Behavioral: Sedentary time breaks every 15 minutes
- 60-15 (Experimental): Sitting for 8 hours interrupted by 3 min of light intensity walking (LIW, 3.2 km/h) breaks every 60 min and 15 min
  Interventions: Behavioral: Sedentary time breaks either every 60 minutes; Behavioral: Sedentary time breaks every 15 minutes
- 30-60 min (Experimental): Sitting for 8 hours interrupted by 3 min of light intensity walking (LIW, 3.2 km/h) breaks every 30 min and 60 min
  Interventions: Behavioral: Sedentary time breaks either every 60 minutes; Behavioral: Sedentary time breaks either every 30 minutes
- 15-30 min (Experimental): Sitting for 8 hours interrupted by 3 min of light intensity walking (LIW, 3.2 km/h) breaks every 15 min and 30 min
  Interventions: Behavioral: Sedentary time breaks either every 30 minutes; Behavioral: Sedentary time breaks every 15 minutes

INTERVENTIONS:
Behavioral: Sedentary time breaks either every 60 minutes — Sitting for 8 hours interrupted by 3 min of light intensity walking (LIW, 3.2 km/h) breaks every 60 min
  Other Names: Sitting for 8 hours interrupted by 3 min of light intensity walking (LIW, 3.2 km/h) breaks either every
  Arms: 15-60 min; 30-60 min; 60-15; 60-30 min
Behavioral: Sedentary time breaks either every 30 minutes — Sitting for 8 hours interrupted by 3 min of light intensity walking (LIW, 3.2 km/h) breaks every 30 min
  Other Names: Sitting for 8 hours interrupted by 3 min of light intensity walking (LIW, 3.2 km/h) breaks every 30 min
  Arms: 15-30 min; 30-15 min; 30-60 min; 60-30 min
Behavioral: Sedentary time breaks every 15 minutes — Sitting for 8 hours interrupted by 3 min of light intensity walking (LIW, 3.2 km/h) breaks every 15 min
  Other Names: Sitting for 8 hours interrupted by 3 min of light intensity walking (LIW, 3.2 km/h) breaks either every 15 minutes
  Arms: 15-30 min; 15-60 min; 30-15 min; 60-15

SUMMARY:
Type-2 diabetes, a common non-infectious disease, is the result of impaired insulin function and insulin production in the body. In type-2 diabetic patients, postprandial glucose control, lipid control and reduction of insulin resistance are crucial to deter the development of diabetes related complications (e.g. retinopathy, nephropathy, neuropathy and cardiovascular diseases), pancreatic β cells failure, morbidity and mortality. Currently, diet, exercise and standard oral medicines are used to treat type-2 diabetes. However, providing the most effective treatment to control postprandial glucose and lipid; and to preserve the pancreatic β cells is challenging because poor metabolic profiles are still detected in type-2 diabetic patients. Therefore, understanding the factors influencing the poor metabolic profiles and adjunct therapy to manage type-2 diabetes are really important to tackle this disease.

In modern society, people are spending most of their waking time in sedentary behaviour, which is primarily prolonged sitting. Prolonged sedentary time is associated with increased postprandial glucose, lipid and insulin resistance. In contrast, frequent interruption of prolonged sitting with short light activity break reduces postprandial glucose, triglyceride cholesterol and insulin resistance. However, how frequently patients should interrupt sitting, potential longer-term effect of short activity break on reduction of postprandial glucose, triglyceride cholesterol and insulin resistance, and the knowledge, beliefs and experiences on the use of technology to decrease sedentary behaviour and improve glycaemic control are not investigated in type-2 diabetic patients. Therefore, it would be relevant to investigate this to prove the therapeutic role of frequent short activity break in sedentary time in the management of type-2 diabetes.

Primary Research Objective:

1. To investigate the dose-response effect of frequency/number of light intensity walking breaks of sitting on postprandial glucose, insulin, C-peptide and triglyceride cholesterol level.
2. To investigate the potential longer-term effect of light intensity walking breaks of sitting on glucose control using 24-h glucose data.

Secondary Research Objectives: The secondary objectives are

1. To obtain data to inform the development of a future feasibility trial investigating the feasibility, compliance, adherence and longer-term effect of different frequencies of light intensity walking breaks in sitting time on glycaemic excursions in free-living.
2. To explore the knowledge, beliefs and experiences of those with Type 2 diabetes on the use of technology to decrease sedentary behaviour and improve glycaemic control, that could be used in the feasibility trial

DETAILED DESCRIPTION:
Overall Study Design:

The study is a three-treatments, two-periods balanced incomplete block trial. Participants will be randomized in blocks completing to two of the three treatment conditions (lab interventions A, B and C below), in different sequence. The three treatment conditions are;

* Intervention A: Sitting for 8 hours interrupted by 3 min of light intensity walking (LIW, 3.2 km/h) breaks every 60 min
* Intervention B: Sitting for 8 hours interrupted by 3 min of light intensity walking (LIW, 3.2 km/h) breaks every 30 min
* Intervention C: Sitting for 8 hours interrupted by 3 min of light intensity walking (LIW, 3.2 km/h) breaks every 15 min There will be 5 days of washout period between each intervention. Each participant will complete two of three treatment conditions within 15 days of experimental period (4 days of pre monitoring period - 1 day of lab intervention - 5 days of washout period - 1 day of lab intervention - 4 days of post monitoring period).

The participants will wear the Abbot FreeStyle Libre continuous glucose monitoring device and the activPAL (activity monitor) throughout the 15 days of experimental period.

Pre-monitoring period: On day 1 of the experimental period, participants will be requested to come to the Diabetes Clinic (Ayr hospital). Baseline anthropometric data (e.g. age, gender, height, weight and body mass index) and drug history will also be recorded by the researcher. The participant will then be fitted with the Abbot FreeStyle Libre continuous glucose monitoring device (sensor) and the activPAL, activity monitor. We will also provide the participant with 24 h diet recall forms so that they can record their daily food intake throughout study period (15 days). After that the participants will return home, instructed to scan their blood glucose every 8 h using the FreeStyle Libre reader they will be supplied with, to record daily food intake, to refrain from smoking, alcohol, caffeine and moderate to vigorous physical activity throughout the experimental period, and to come back on day 5.

Lab intervention 1: On day 5 of the experimental period (intervention day), participants will arrive at the Diabetes Clinic (Ayr hospital) at 08:00 h after an overnight fast. Prof. A Collier (Chief Investigator) and the researchers will meet with participants at the reception. The participant will be seated from 08:00 h to 09:00 h, to achieve a physiological steady state, in the consulting room (private room). During this period, an intravenous catheter will be inserted into an antecubital vein for hourly blood collection by clinicians (two clinical teaching fellows) and, the researcher will explain the procedure and offer choices of entertainment (e.g. TV, DVD, Books and Magazine). At 09:00 h, the participant will consume a standardised meal/breakfast (weetabix 52 grams plus 250ml full fat milk = 50grams of carbohydrates or cornflakes 45.4 grams plus 250ml full fat milk = 50 grams of carbohydrates). After that the participant will perform 3 min of light intensity walking (LIW) either every 60 minutes (Intervention A), 30 minutes (Intervention B) or 15 minutes (Intervention C) of sitting on a motorised treadmill with a pace of 3.2 km/h. This sequence will continue until the end of the intervention (16:00 h). Timing will be done by the researcher who will be in the room with participant. The researcher will instruct the participant to stand and walk on the treadmill as per the timing of the specific condition. The participant will be guided to the treadmill which will be started slowly by the researcher and this will increase to 3.2 km/h. At the end of the walking period, the researcher will slowly decrease the speed until the participant comes to steady standing. The participant will then be instructed to resume the sitting position. Every hour the clinicians (two clinical teaching fellows) will collect 12 ml of blood samples from patients through the inserted catheter. This sequence will be repeated until the condition is completed.

At 12:36 h, the participant will be served a standardised lunch (sandwich x 2 slices thick bread 40 grams carbohydrates, yogurt 14-16 grams carbohydrates, crisps 25 gram multipack bag 13-15 grams carbohydrates) during that sitting period. At the end of the intervention the intravenous catheter will be removed by clinicians (two clinical teaching fellows). A standardised dinner (sandwich x 2 slices thick bread 40 grams carbohydrates, yogurt 14-16 grams carbohydrates, crisps 25 gram multipack bag 13-15 grams carbohydrates) will also be provided, and participants will be instructed to have this dinner at 17:00 h at home. Participants will be instructed to avoid having any other food on that day apart from the standardised dinner provided.

Washout period: There will be 5 days of washout period between two treatment conditions (interventions A, B and C). The chief investigator and the researchers will stay in touch with the participants during this period so that they can remind the participants to come back and to perform another lab intervention after 5 days. The chief investigator and the researchers will use the mode of communication which is the most convenient to the participant (phone or email) to contact them and schedule visits.

Lab intervention 2: On day 11 of experimental period, the participant will come back and arrive at the Diabetes Clinic (Ayr hospital) at 08:00 h after an overnight fast to perform the lab intervention 2. Every procedure of the lab intervention 2 will be the same as the lab intervention 1 except for performing another of three treatment conditions, which was not performed during lab intervention 1.

Post-monitoring period: Physical activity and continuous glucose monitoring will continue for four days, from day 12 to day 15 of experimental period, after the lab intervention 2. This will be regarded as post-monitoring period. During this period participants will also be reminded to avoid caffeine, alcohol, smoking and moderate to vigorous physical activity. On day 15, participants will report back to the laboratory (Diabetes Clinic at Ayr Hospital) in the morning for removal of the Abbot FreeStyle Libre continuous glucose monitoring device and the activPAL. After that, participants will be thanked and they will return home. This will be the end of experimental period for each participant.

Qualitative investigations: During the second laboratory intervention, the participants will be asked to take part in a one to one interview. The interview will be semi-structured and focus on the participant's views and experiences of the use of mobile-based technology in Type 2 diabetes management. During the interview, the participant will be shown a variety of mobile-based technology that is currently available including wearable technology and mobile/tablet apps.

The interview questions will cover the participant's knowledge of sedentary behaviour, their views on regular breaks in sedentary behaviour, the use of technology in promoting breaks in sedentary behaviour and their experiences of using technology to increase their breaks in sedentary behaviour to improve their glycaemic control. All interviews will be tape recorded with the participants' permission and, due to the flexible nature of the process and individual responses of the participants, it is anticipated that each interview will last 1 hour.

Research questions for qualitative investigations:

1. Are people with Type 2 diabetes aware of the health benefits of low levels of sedentary behaviour?
2. How often do those with Type 2 diabetes think they could feasibly break their sedentary behaviour?
3. Are they aware of or ever used mobile-based technology to improve their health?
4. What are the views and experiences of those with Type 2 diabetes on using mobile-based technology as a method of improving their glycaemic control?

Subject Information and Consent:

Type-2 diabetic patients (N=24) will be used in this study. Potential participants will be given information about the study. If the potential participant is willing, Prof. A Collier and the researchers will send the study information pack and consent form to the participant. The potential participant will also be given oral explanations about the procedures of the study by Prof. A Collier and the researchers. A week later, the clinic will contact the potential participant again to ascertain if they have received the pack or if they have any further question. At that point, the clinic will ask if the potential participant is willing to enter the study and if so, request that they return the consent form. An appointment for visit one will then be made. A schedule of appointment for the whole study will be agreed with the participant and given in writing to the participants. The participants will be asked about how they want to be contacted for reminders. In addition, the participant will be given a contact number to call the researcher if they have any question or queries at any stages. Prof A. Collier and the researchers will also send a letter to the patient's GP explaining detail of study.

Data Collection:

The glucose excursions and physical activity level of the participants will be monitored by Abbot FreeStyle Libre continuous glucose monitoring device and activPAL (activity monitor) throughout study period. Moreover, hourly venous blood will also be taken from the participants during each lab interventions to assess the postprandial glucose, insulin, C-peptide and triglyceride cholesterol levels.

Data Management:

In accordance with the Data Protection Act 1998, all subject data will be anonymised and each patient will be given a unique research number. The study data (consent, patient demographics, laboratory results, details of intervention) will be stored in a locked filing cabinet in the Chief Investigator's office which is also locked. Electronic data will be stored on the NHS server on an access database. Memory sticks will not be used to store data. Each patient will be given a unique identifier. All study data will be anonymised and only the members of the research team will have access.

The audio files from the qualitative investigation will be transferred immediately to a password protected computer in the Graham Hills building, University of Strathclyde. The audio files will be deleted from the recording device as soon as the files have been transferred to the University password protected computer. The interviews will be transcribed, these transcriptions will be anonymised (i.e. using participants' unique identifier), hard copies of the anonymised transcriptions will be stored in a locked filing cabinet, and electronic copies of the anonymised transcriptions will be stored on a password protected computer based in the Graham Hills building, University of Strathclyde.

Data Analysis:

If the data is normally distributed, differences between variables (postprandial glucose, insulin, C-peptide, triglyceride and 24 h glucose) of intervention groups will be analysed using multiple mixed-effects linear regression method allowing for repeated measurements from the same individuals. Treatment condition and the participant will be regarded as a fixed factor and a random factor respectively. Prior to analysis all outcomes will be tested for assumption of normality. In case of non-normality, data transformation will be applied and if this is not satisfactory the analysis will be carried out using non-parametric equivalent techniques. Models will be corrected for age, gender, physical activity and baseline measurements, diabetes history, drug intake and diet.

Reporting for Adverse Events:

All adverse events will be recorded and reported. Subjects will be specifically asked about adverse events. All events will be recorded by the investigator in an Adverse Event form and each event will be recorded separately. The research team do not anticipate any adverse AEs. However, if there is an AE the research team will report the incident to NHS Ayrshire and Arran Health Board's R&D Office within 24 hours and this will be followed up as per the R&D policies and procedures.

Reporting for Serious Adverse Events or Suspected Unexpected Serious Adverse Events:

The research team does not anticipate any serious adverse events (SAE) or suspected unexpected serious adverse events (SUSAEs). However, if any of these occur then the research team will report the incident to NHS Ayrshire & Arran R&D office within 24 hours and this will be followed up as per R&D policies and procedures.

Change Management:

The Investigator will not deviate from the protocol without agreement from the Prof. A Collier (Chief Investigator), and REC and R&D approval, except if necessary to remove an apparent immediate hazard to the participant. In the event that this is necessary, the nature of and reasons for the deviation should be recorded. If this necessitates a subsequent protocol amendment this should be submitted in writing to the appropriate REC and Research and Development office for review and approval if appropriate.

Sample Size Assessment:

Based on available data from laboratory studies, it is estimated that a sample size of 24 in a three-treatment two-period balanced incomplete block design should be sufficient to detect the significant effect of frequent short bouts of light intensity activity breaks on postprandial glucose reduction with a statistical power of 80% and 95% confidence.

Procedures for Accounting for Missing, Unused and Spurious data:

The trial will be analysed both as 'intention to treat' and 'per protocol'. In the intention to treat analysis missing data will be replaced with baseline data. In the 'per protocol' analysis participants with missing data will not be considered.

Statistical Analysis Plan:

If the data is normally distributed, differences between variables (postprandial glucose, insulin, C-peptide, triglyceride and 24 h glucose) of intervention groups will be analysed using multiple mixed-effects linear regression method allowing for repeated measurements from the same individuals. Treatment condition and the participant will be regarded as a fixed factor and a random factor respectively. Prior to analysis all outcomes will be tested for assumption of normality. In case of non-normality, data transformation will be applied and if this is not satisfactory the analysis will be carried out using non-parametric equivalent techniques. Models will be corrected for age, gender, physical activity and baseline measurements, diabetes history, drug intake and diet.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with type 2 diabetes for less than 10 years
* Individuals aged 35-60 years
* Individuals receiving metformin or diet control
* Non-smokers
* Overweight and obese individuals (BMI 25-35 kg/m2)
* Individuals with an HbA1c between >7%
* Individuals with BP below 160/90mmHg

Exclusion Criteria:

* Individuals unable or unwilling to consent
* Individuals under the age of 35 years and over the age of 60 years at study enrolment
* Patients on sulphonylurea or other oral hypoglycaemic drugs therapy except metformin
* Individuals with hepatic or renal dysfunction
* Individuals with body mass index greater than 35
* Individuals suffering from cancer, cardiovascular diseases, cirrhosis, hepatitis and renal disease
* Pregnant Individuals
* Individuals who smoke
* Individuals who are alcohol and drug abusers
* Individuals with a blood pressure ≥160/90mmHg
* Individuals diagnosed with anaemia (Hb<12g/dl in women and <13 g/dl in men)
* Individuals taking medicines which can interfere with the glucose metabolism (e.g. anticoagulants, oral contraceptives, steroid, thiazide, β-blocker, NSAID, anti-fungal, hormonal therapy, psychotropic drugs)
* Individual taking drugs for glycaemic control in excess of standard care highlighted by the SIGN guideline 116.

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-01 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Postprandial glucose excursions measured with Area under curve | 8 hours
  Dose-response relationship between frequencies of short light activity breaks in sedentary time and postprandial glucose excursions

SECONDARY OUTCOMES:
24 hours glucose profile measured with continuous glucose monitor LifeStyle Libre | 24 hours
  The effect of interruption of sedentary time with frequent short activity break on 24 hr glucose profile, insulin, C-peptide and triglyceride cholesterol levels will be assessed during each intervention. Then knowledge, beliefs and experiences of the type-2 diabetic patients on the use of technology to decrease sedentary behaviour and improve glycaemic control will be assessed.
Insulin, C-peptide and triglyceride cholesterol plasma level during the intervention measured with Area under curve | 8 hours
  The effect of interruption of sedentary time with frequent short activity break on 24 hr glucose profile, insulin, C-peptide and triglyceride cholesterol levels will be assessed during each intervention. Then knowledge, beliefs and experiences of the type-2 diabetic patients on the use of technology to decrease sedentary behaviour and improve glycaemic control will be assessed.
Qualitative exploration of the knowledge, beliefs and experiences of those with type 2 diabetes on the use of technology to decrease sedentary behaviour and improve glycaemic control | 1 hour
  The effect of interruption of sedentary time with frequent short activity break on 24 hr glucose profile, insulin, C-peptide and triglyceride cholesterol levels will be assessed during each intervention. Then knowledge, beliefs and experiences of the type-2 diabetic patients on the use of technology to decrease sedentary behaviour and improve glycaemic control will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Collier,, MBchb, Principal Investigator — Glasgow Caledonian University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chastin SF, Egerton T, Leask C, Stamatakis E. Meta-analysis of the relationship between breaks in sedentary behavior and cardiometabolic health. Obesity (Silver Spring). 2015 Sep;23(9):1800-10. doi: 10.1002/oby.21180. PMID 26308477
- [Background] Cooper AR, Sebire S, Montgomery AA, Peters TJ, Sharp DJ, Jackson N, Fitzsimons K, Dayan CM, Andrews RC. Sedentary time, breaks in sedentary time and metabolic variables in people with newly diagnosed type 2 diabetes. Diabetologia. 2012 Mar;55(3):589-99. doi: 10.1007/s00125-011-2408-x. Epub 2011 Dec 14. PMID 22167127
- [Background] Dempsey, P.C., Owen, N., Larsen, R., Straznicky, N., Cohen, Neale., FACSM, B.B., Kingwell, B.A., Dunstan, D.W., Baker IDI Heart and Diabetes Institute, Melbourne, Australia., Department of Health and Exercise Science, Colorado State University, Fort Collins, Colorado, USA. 2015. Interrupting Prolonged Sitting: A Potential Therapeutic Tool in the Management of Type 2 Diabetes
- [Background] Dunstan DW, Kingwell BA, Larsen R, Healy GN, Cerin E, Hamilton MT, Shaw JE, Bertovic DA, Zimmet PZ, Salmon J, Owen N. Breaking up prolonged sitting reduces postprandial glucose and insulin responses. Diabetes Care. 2012 May;35(5):976-83. doi: 10.2337/dc11-1931. Epub 2012 Feb 28. PMID 22374636
- [Background] Healy GN, Dunstan DW, Salmon J, Cerin E, Shaw JE, Zimmet PZ, Owen N. Breaks in sedentary time: beneficial associations with metabolic risk. Diabetes Care. 2008 Apr;31(4):661-6. doi: 10.2337/dc07-2046. Epub 2008 Feb 5. PMID 18252901
- [Background] Henson J, Yates T, Biddle SJ, Edwardson CL, Khunti K, Wilmot EG, Gray LJ, Gorely T, Nimmo MA, Davies MJ. Associations of objectively measured sedentary behaviour and physical activity with markers of cardiometabolic health. Diabetologia. 2013 May;56(5):1012-20. doi: 10.1007/s00125-013-2845-9. Epub 2013 Mar 1. PMID 23456209
- [Background] Latouche C, Jowett JB, Carey AL, Bertovic DA, Owen N, Dunstan DW, Kingwell BA. Effects of breaking up prolonged sitting on skeletal muscle gene expression. J Appl Physiol (1985). 2013 Feb 15;114(4):453-60. doi: 10.1152/japplphysiol.00978.2012. Epub 2012 Dec 27. PMID 23271697
- [Background] Peddie MC, Bone JL, Rehrer NJ, Skeaff CM, Gray AR, Perry TL. Breaking prolonged sitting reduces postprandial glycemia in healthy, normal-weight adults: a randomized crossover trial. Am J Clin Nutr. 2013 Aug;98(2):358-66. doi: 10.3945/ajcn.112.051763. Epub 2013 Jun 26. PMID 23803893
- [Derived] Paing AC, McMillan KA, Kirk AF, Collier A, Hewitt A, Chastin SFM. Dose-response between frequency of interruption of sedentary time and fasting glucose, the dawn phenomenon and night-time glucose in Type 2 diabetes. Diabet Med. 2019 Mar;36(3):376-382. doi: 10.1111/dme.13829. Epub 2018 Oct 12. PMID 30264906